CLINICAL TRIAL: NCT03766035
Title: Cholangioscopy in Primary Sclerosing Cholangitis (PSC)
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E7136
Record Dates: First submitted 2018-11-08; First posted 2018-12-05 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
Keywords: per oral cholangioscopy; PSC; cholangiocarcinoma; primary sclerosing cholangitis; ERCP
MeSH Terms: conditions — Cholangitis, Sclerosing; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Consented, enrolled PSC patients undergoing ERCP + SpyGlass: Patients with PSC who have been consented and enrolled in the study will undergo ERCP with the addition of SpyGlass as indicated by their treating physician.
  Interventions: Device: SpyGlass DS I - II

INTERVENTIONS:
Device: SpyGlass DS I - II — The SpyScope™ DS Access and Delivery Catheter (SpyScope™ DS Catheter) is a sterile, single-use endoscope that enables access and delivery of accessories to targeted pancreaticobiliary anatomy and displays live video when connected to a Spy Glass DS Digital Controller.

SUMMARY:
To demonstrate the clinical utility of the addition of per oral cholangioscopy (POCS) to standard endoscopic retrograde cholangiopancreatography (ERCP) with brushing cytology for diagnosis and early detection of cholangiocarcinoma in patients diagnosed with primary sclerosing cholangitis (PSC).

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the clinical utility of the addition of per oral cholangioscopy (POCS) to standard ERCP with brushing cytology for diagnosis and early detection of cholangiocarcinoma in patients diagnosed with primary sclerosing cholangitis (PSC).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of PSC
2. Clinical indication for ERCP per local standard of practice, such as suspicion of potential malignancy based on worsening cholestatic values or clinical presentation (such as itching, cholangitis) or new biliary stricture on trans-abdominal imaging (MRI/MRCP, US or CT) or suspicious cytology
3. Diameter of bile ducts deemed sufficient to accommodate the cholangioscopy system based on imaging performed prior to scheduled ERCP
4. Written informed consent from patient to participate in the study, including compliance with study procedures.

Exclusion Criteria:

1. Contraindication for an ERCP or POCS
2. History of liver transplantation
3. Mass/metastasis extrinsic to the bile duct identifiable on diagnostic imaging
4. History of iatrogenic bile duct trauma, including biliary surgery within 6 months of enrollment
5. INR > 1.5 or platelets count < 50,000
6. Age < 18 years
7. Pregnant women or women trying to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with PSC
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of POCS visualization for Early Detection of Cholangiocarcinoma | 12 months
  Diagnostic accuracy of POCS visualization for cholangiocarcinoma evaluated clinically at 12 months after initial POCS procedure by clinical presentation.
POCS-guided Biopsy for Early Detection of Cholangiocarcinoma | 12 months
  Diagnostic accuracy for POCS-guided Biopsy for cholangiocarcinoma evaluated on pathology at 12 months after initial POCS procedure.

SECONDARY OUTCOMES:
Technical Success - Ability to advance the scope. | Baseline
  Ability to advance the cholangioscope to the target stricture, ability to visualize the stricture and ability to obtain a tissue sample with Spy Bite where applicable.
Rate of Adverse Events | From index through study completion, an average of one year
  Serious adverse events from initial POCS procedure until end of follow-up.
Proportion of patients identified for repeat procedure. | During index procedure
  Proportion of patients identified for repeat procedure considering the addition of Spy Glass DS visualization and Spy Bite biopsy at Index compared to the proportion identified for repeat procedure without consideration of Spy Glass DS visualization and Spy Bite biopsy at Index.
Correspondence of Biopsies | From index through study completion, an average of one year
  Correlation between histopathology of Spy Bite biopsies collected during the initial POCS procedure and final diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Eksteen, MD, PhD, Principal Investigator — Aspen Woods Clinic; Douglas Adler, MD, Principal Investigator — University of Utah Hospital and Clinic; Lars Aabakken, MD, PhD, Principal Investigator — Rikshospitalet Oslo University Hospital; Cyriel Ponsioen, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Sooraj Tejaswi, MD, PhD, Principal Investigator — Sutter Davis Hospital; Christopher Bowlus, MD, PhD, Principal Investigator — UC Davis Health
Locations (6):
- United States (3):
  - Sutter Davis Hospital, Davis, California
  - UC Davis Health, Sacramento, California
  - University of Utah Hospital and Clinic, Salt Lake City, Utah
- Aspen Woods Clinic, Calgary, Alberta, Canada
- Academic Medical Center, Amsterdam-Zuidoost, Netherlands
- Rikshospitalet University Hospital, Oslo, Norway